CLINICAL TRIAL: NCT04293497
Title: Clinical Validation of a New Immunochemistry Method Using Antibody of Methionyl-tRNA synthetase1(MARS1) in the Pancreatic Cancer Cell; Multicenter Prospective Study
Brief Title: Development of a New Immunochemistry Method Using Antibodies of Proteins Related Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung III Jang, Associate professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2019-0410
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The conventional staining method and new staining method will be performed in cytology specimens obtained from same patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pancreatic Cancer (Experimental): This arm includes patients with pancreatic cancer. Cytology specimens will be obtained with endoscopic ultrasound-guided fine-needle aspiration in patients with pancreatic cancer. Cytology staining will be performed in the cytology specimens.
  Interventions: Diagnostic Test: Cytology staining

INTERVENTIONS:
Diagnostic Test: Cytology staining — Two staining will be performed in cytology specimens obtained from same patient. The cytology specimen will be obtained using endoscopic ultrasound-guided fine needle aspiration. Three types of slides (direct smear, thinprep, surepath) are prepared for staining.
  1. conventional cytology staining method
  2. new cytology staining method using antibody of methionyl-tRNA synthetase 1

SUMMARY:
Identifying the malignancy of pancreatic mass using endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) is important for treatment decision-making and prognosis prediction. The sensitivity of EUS-FNA cytology specimens based on Papanicolaou (Pap) staining is low, which hampers accurate diagnosis of pancreatic mass. We assessed the diagnostic value of immunohistochemical (IHC) and immunofluorescence (IF) staining for methionyl-tRNA synthetase 1 (MARS1).

DETAILED DESCRIPTION:
BACKGROUND / AIMS: The sensitivity of endoscopic ultrasound-guided aspiration cytology used to distinguish the pancreatic mass is low and clinical usefulness is not secured. The aim of this study was to evaluate clinical efficacy of a new differential staining method for cytology which is difficult to differentiate by the conventional staining method using pancreatic cancer related protein expressed only in pancreatic cancer.

Hypothesis: The statistical significance between conventional staining method and MARS1 staining in the pancreatic cancer cells collected by endoscopic ultrasound-guided aspiration will be compared to prove the usefulness of the new staining method.

Clinical study design: The expression of MARS1 in the pancreatic cancer cell line obtained by endoscopic ultrasound in patients suspected of having pancreatic cancer using Immunofluorescence or immunohistochemistry staining will be performed to differentiate the presence of the tumor. The sensitivity and specificity of the new staining method will be compared with the conventional staining method and its usefulness be confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pancreatic cancer confirmed by imaging (CT, MRI, PET-CT)
2. Patients with pancreatic cancer diagnosed using cytology by endoscopic ultrasound
3. Patients who underwent surgical treatment with pancreatic cancer

Exclusion Criteria:

1. Minors under the age of 19, vulnerable subjects such as illiteracy
2. Excludes necrotic specimens
3. Samples with non-diagnostic cytology results and insufficient cells for further evaluation
4. Samples classified as neoplastic (benign or other)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
The comparison of sensitivity between conventional staining method and new staining method | 1 year
  The sensitivity of new staining method will be compared with the conventional Pap staining of endoscopic ultrasound-guided fine-needle aspiration cytology

SECONDARY OUTCOMES:
The evaluation of correlation index of staining at three type slides | 1 year
  The correlation index of the new staining method will be evaluated at three type slides such as Thinprep, Surepath, and Direct smear.

CONTACTS AND LOCATIONS:
Overall Officials: Sung III Jang, MD, PhD, Principal Investigator — Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (4):
- South Korea (4):
  - CHA Bundang Medical Center, Seongnam, Bundang-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - In Ha University Hospital, Incheon, Jung-gu
  - Soon Chun Hyang University Hospital, Cheonan, Cheonan, Namdong-gu

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the following individual participant data with other researchers during study period.
  Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR), Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: Primary investigator Sub primary investigator